CLINICAL TRIAL: NCT06687772
Title: Safety and Feasibility Study for CNS-Relapse Prevention in High-Risk Diffuse Large B-cell Lymphoma With Thiotepa-based Autologous Stem Cell Transplant (CNS-PHLAT)
Brief Title: CNS-Relapse Prevention in High-Risk Diffuse Large B-cell Lymphoma With Thiotepa-based Autologous Stem Cell Transplant
Acronym: CNS-PHLAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202411136
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; Autologous stem cell transplant; CNS lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Thiotepa; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Anthracycline-based induction chemotherapy + ASCT + Thiotepa + Carmustine (Experimental): * Patients should receive induction treatment with anthracycline-based chemotherapy regimen per standard of care. Between the end of induction Cycle #2 and the end of induction Cycle #4, a PET/CT scan should be performed to assess response. If there are no signs of progressive disease and the treating physician recommends patient is eligible for ASCT, patients should be consented with the treatment consent. Treatment with thiotepa and carmustine may not take place prior to this second patient consent. Within 3 weeks after the end of the final cycle of induction, a PET-/CT scan should be performed to assessconfirm treatment response and eligibility for ASCT.
  * After signing the treatment consent and confirming complete response (CR) following induction therapy, patients will begin conditioning with thiotepa (days -5 and -4) and carmustine (day -6), followed by ASCT on day 0.
  Interventions: Drug: Thiotepa; Drug: Carmustine; Procedure: Autologous Stem Cell Transplant; Drug: Anthracycline-based induction chemotherapy

INTERVENTIONS:
Drug: Thiotepa — Thiotepa will be given intravenously twice daily on Days -5 and -4 over 120 minutes at a dose of 5 mg/kg.
Drug: Carmustine — Carmustine will be given intravenously on Day -6 over 120 minutes at a dose of 400 mg/m^2.
Procedure: Autologous Stem Cell Transplant — Infusion of autologous peripheral blood stem cells on Day 0.
  Other Names: ASCT
Drug: Anthracycline-based induction chemotherapy — Standard of care, not dictated by protocol.

SUMMARY:
A serious consequence of systemic diffuse large B-cell lymphoma (DLBCL) is secondary central nervous system (CNS) relapse, which occurs in approximately 5% of all patients. Many CNS relapses occur within the first year after completion of frontline treatment and are associated with significantly increased mortality; thus, it is important to tailor frontline treatment to provide prophylaxis against CNS relapse in those patients who are determined to be high-risk.

Autologous stem cell transplantation (ASCT) is standard of care for patients with DLBCL who relapse one year or more after first remission, and it has been shown to improve progression-free survival for patients with primary CNS lymphoma.

The four-drug BEAM regimen (carmustine, etoposide, cytarabine, and melphalan) is the preferred conditioning regimen for DLBCL patients undergoing ASCT; however, patients with primary CNS lymphoma receive thiotepa plus carmustine as their conditioning regimen due to its better CNS penetration.

This study tests the hypothesis that consolidation thiotepa/carmustine ASCT in first complete remission will reduce the risk of CNS relapse in transplant-eligible patients with DLBCL with no prior CNS disease at high risk of secondary CNS recurrence.

ELIGIBILITY:
Screening Inclusion Criteria:

* Newly diagnosed diffuse large B-cell lymphoma, large B-cell lymphoma transformed from underlying indolent lymphoma, or high-grade B-cell lymphoma. Patients with secondary CNS lymphoma are eligible. Patients with Richter's transformation are NOT eligible.
* At high risk for CNS relapse prior to start of induction as defined by at least one of the criteria below:

  * CNS-IPI ≥ 4
  * Kidney or adrenal involvement
  * Testicular involvement
  * Breast involvement
  * Ovarian involvement
  * Uterine involvement
  * Skin involvement
  * Double hit lymphoma as defined by containing translocations of MYC gene together with rearrangement of BCL2 and/or BCL6.
  * Bone marrow involvement
  * Myocardium involvement
  * CNS adjacent
  * Secondary CNS involvement
* Intend to receive a full course of curative-intent anthracycline-based induction treatment and has not yet received more than 2 cycles at the time of screening. Can receive induction chemotherapy outside of Siteman if still compliant with study eligibility, laboratory studies, lumbar punctures, imaging, and other events.
* Ages 18 to 75.
* Ability to understand and willingness to sign an IRB-approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants if patient is otherwise unable to sign for themselves or unable to understand consent document.

Treatment Eligibility Criteria:

* Currently undergoing anthracycline-based induction treatment. Dose modifications and/or delays during induction therapy may be made at the discretion of the treating physician and will not affect eligibility for continuation in the study.
* ECOG performance status ≤ 2.
* PET/CT assessment performed between the end of induction Cycle #2 and end of induction Cycle #4 demonstrates no evidence of progressive disease, and patient is eligible for autologous stem cell transplant as determined by the treating physician.
* Has signed treatment consent form following mid-induction PET/CT and prior to conditioning treatment with thiotepa/carmustine.
* Thiotepa and carmustine can cause fetal harm when administered to a pregnant person. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study treatment, and for 6 months following receipt of thiotepa and/or carmustine (for women) and 12 months following receipt of thiotepa and/or carmustine (or 3 months following receipt of carmustine if discontinuing before thiotepa) (for men). Should a woman become pregnant or suspect she is pregnant during treatment or within 6 months of the last dose of either thiotepa or carmustine or should a man suspect he has fathered a child, s/he must inform the treating physician immediately.

Exclusion Criteria (applies at both screening and treatment)

* Relapsed or refractory diffuse large B-cell lymphoma or high-grade B-cell lymphoma. Prior treatment for underlying indolent lymphoma is permitted.
* Diagnosis of primary CNS lymphoma.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen as determined by the PI. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to thiotepa, carmustine, or other agents used in the study.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days prior to start of induction (for people enrolling prior to induction) or within 7 days of enrollment (for people enrolling after the start of induction).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treatment | Through completion of treatment (estimated to be 6 months)
  - The treatment (thiotepa/carmustine conditioning and ASCT) will be considered feasible if > 50% of enrolled patients meet the following criteria:
  * Achieve CR at the end of induction chemotherapy
  * Remain eligible for ASCT
  * Collect sufficient stem cells for ASCT (CD34+ cell goal ≥2 x 10^6/kg)
  * Complete thiotepa/carmustine chemotherapy and undergo ASCT

SECONDARY OUTCOMES:
Rate of selected transplant-related grade 3-5 adverse events | From start of study treatment through day 30 after transplant (estimated to be 7 months)
Rate of CNS relapse | At 2 years post-thiotepa/carmustine conditioning and ASCT (estimated to be 2.5 years)
Progression-free survival (PFS) | At 2 years post-thiotepa/carmustine conditioning and ASCT (estimated to be 2.5 years)
Overall survival (OS) | At 2 years post-thiotepa/carmustine conditioning and ASCT (estimated to be 2.5 years)
Non-relapse mortality | At 2 years post-thiotepa/carmustine conditioning and ASCT (estimated to be 2.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda F Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu